CLINICAL TRIAL: NCT04358224
Title: The Utility of Functionally Relevant Signature Genes in Assessing the Clinical Outcomes of Dupilumab Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jonathan A. Bernstein, MD (Other)
Responsible Party: Sponsor-Investigator, Jonathan A. Bernstein, MD, principal investigator, Bernstein Clinical Research Center
Organization: Bernstein Clinical Research Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R668-AD-1830
Record Dates: First submitted 2020-04-14; First posted 2020-04-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- open-label (Other): open-label
  Interventions: Biological: Dupilumab Prefilled Syringe

INTERVENTIONS:
Biological: Dupilumab Prefilled Syringe — open-label
  Other Names: dupixent

SUMMARY:
The utility of functionally relevant signature genes in assessing the clinical outcomes of dupilumab treatment in the adult onset atopic dermatitis

DETAILED DESCRIPTION:
The study consists of 9 visits. Duplimab will used in the treatment of adult onset atopic dermatitis. Qualified subjects will receive 5 dupilumab open-label injections. Skin biopsies/ skin strips will be obtained at the beginning and the end of treatment. TARC and IgE levels will be obtained at the beginning and end of treatment. Subjects will complete daily diaries assessing atopic dermatitis symptoms. Patient reported out comes will be completed at each visit

ELIGIBILITY:
Inclusion Criteria:

* history of adult onset atopic dermatitis

Exclusion Criteria:

-

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to correlate cutaneous transcriptomes with before and after Dupilumab treatment outcomes in patients who meet the clinical diagnostic criteria for adult onset AD. | after 6 months
  Data will be analyzed from skin punch biopsies from active skin lesions and uninvolved skin samples before and after treatment

SECONDARY OUTCOMES:
To investigate possible influence of Dupilumab on serologic protein biomarkers in patients with adult onset AD | after 6 months
  Total IgE, TARC and eotaxin will be compared pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bernstein, Principal Investigator — Bernstein Clinial Research Center
Locations (1):
- Bernstein Clinical Research Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
to be determined
Supporting Information: Study Protocol, SAP, CSR
Time Frame: at end of trial
Access Criteria: to be determined